CLINICAL TRIAL: NCT07286877
Title: Enhanced Ward-Round Frequency With Standardized Communication for Pre-procedural Anxiety in Hospitalized Patients Undergoing Therapeutic Gastrointestinal Endoscopy
Brief Title: Enhanced Ward Rounds and Communication for Pre-procedural Anxiety in GI Endoscopy Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LanZhou University (Other)
Responsible Party: Principal Investigator, Zhaofeng Chen, Clinical Professor, LanZhou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: LDYYczf2025110501
Record Dates: First submitted 2025-11-14; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Anxiety; Depression Disorders; Sleep Wake Disorders; Gastrointestinal Diseases; Preoperative Anxiety
MeSH Terms: conditions — Anxiety Disorders; Sleep Wake Disorders; Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Ward Rounds (4/day) with Standardized Communication (Experimental): In intervention wards/periods, the care team conducts four brief, structured ward-round contacts per day (morning 07:00-09:00, midday 11:00-13:00, afternoon 15:00-17:00, and bedtime 19:00-21:30), each lasting approximately 3-5 minutes. Each contact uses a standardized communication script addressing patient concerns, provides concise procedure-related education, and includes a 2-3 minute relaxation/breathing exercise. For patients undergoing lower GI procedures, a bowel preparation checklist is reviewed and an information card is issued/verified at each contact. Delivery starts at enrollment and continues through 24-48 hours post-procedure or until discharge, whichever comes first. Staff receive standardized training with competency assessment; fidelity is monitored via daily checklists with an adherence target of ≥85%. All usual clinical care remains available at all times.
  Interventions: Behavioral: Enhanced Ward-Round Frequency With Standardized Communication
- Usual Care Ward Rounds (2/day) (Active Comparator): Routine ward rounds twice daily (morning 07:00-09:00 and afternoon 15:00-17:00) according to standard hospital practice, without additional structured rounds, standardized communication scripts, scheduled relaxation exercises, or structured bowel preparation checklists beyond usual patient education. Applied from enrollment through 24-48 hours post-procedure or until discharge, whichever comes first. Clinically necessary additional contacts are permitted and recorded as protocol deviations. All other aspects of care follow standard institutional pathways.
  Interventions: Behavioral: Usual Care Ward Rounds (2/day)

INTERVENTIONS:
Behavioral: Enhanced Ward-Round Frequency With Standardized Communication — In intervention wards/periods, the care team conducts four brief, structured ward-round contacts per day (morning, noon, afternoon, and a bedtime contact not later than 21:30), each lasting approximately 3-5 minutes. Each contact uses a standardized communication script that addresses patient concerns, provides concise procedure-related education, and includes a 2-3 minute relaxation/breathing exercise; for lower GI procedures, a bowel preparation checklist is reviewed and an information card is issued/verified. Delivery starts at enrollment and continues through 24-48 hours post-procedure or until discharge, whichever comes first. Staff receive standardized training; fidelity is monitored via daily checklists with an adherence target of ≥85%. Usual clinical care remains available at all times.
  Other Names: Enhanced Ward Rounds; 4/day Ward Rounds; Standardized Communication Package
  Arms: Enhanced Ward Rounds (4/day) with Standardized Communication
Behavioral: Usual Care Ward Rounds (2/day) — Routine ward rounds twice daily (morning and afternoon) according to standard hospital practice, without additional rounds, the standardized communication script, relaxation exercise, or the structured bowel preparation checklist beyond usual education. Applied from enrollment through 24-48 hours post-procedure or until discharge, whichever comes first. Any clinically necessary deviations are permitted and recorded as protocol deviations; all other aspects of care follow standard pathways.
  Other Names: Usual Care; Standard Practice
  Arms: Usual Care Ward Rounds (2/day)

SUMMARY:
This study tests a new way to help reduce anxiety in hospitalized patients waiting for therapeutic gastrointestinal (GI) endoscopy procedures, like EMR or ESD. Anxiety before these procedures is common and can make preparation harder, increase medication needs, and affect recovery.

We compare standard ward checks (twice a day) to enhanced checks (four times a day) with structured talks and simple relaxation exercises. The goal is to see if the enhanced approach lowers anxiety levels, measured by a standard scale called the Hamilton Anxiety Rating Scale (HAM-A), from baseline to 24 hours before the procedure.

Who can join? Adults (18+) scheduled for inpatient GI endoscopy with at least 2 days hospital stay and mild anxiety. Exclusions include emergencies or severe mental health issues.

The study is done in hospital wards, with groups assigned by ward periods to keep it real-world. Benefits may include less anxiety and better experience; risks are low as it's just more supportive talks. Participation is voluntary with informed consent. Results could improve hospital care routines.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Inpatients scheduled for therapeutic gastrointestinal endoscopy (e.g., ESD/EMR, therapeutic colonoscopy).
3. Able to provide informed consent and complete required assessments.

Exclusion Criteria:

Emergency/immediate endoscopy required.

1. Severe cognitive impairment or psychotic disorder affecting assessments. Isolation/single room preventing protocol implementation.
2. Unable to complete the primary pre-procedure assessment within the 2-4 hour window.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-02-20 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton Anxiety Rating Scale (HAM-A) Score | Baseline and 3 hours (±1 hours) before scheduled endoscopy procedure (assessed up to 14 days after enrollment)
  The Hamilton Anxiety Rating Scale (HAM-A) is a clinician-administered instrument assessing anxiety severity. Total score ranges from 0 to 56 points, with higher scores indicating worse anxiety. Score interpretation: 0-7 = no anxiety, 8-16 = mild anxiety, 17-24 = mild-to-moderate anxiety, 25-30 = moderate-to-severe anxiety, >30 = severe anxiety. Assessed by blinded research assistants using structured interview.

SECONDARY OUTCOMES:
Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) Overall Hospital Rating | At hospital discharge (assessed up to 21 days after enrollment)
  HCAHPS Overall Hospital Rating measures patient satisfaction with hospital care on a scale of 0 to 10, where 0 = worst hospital possible and 10 = best hospital possible. Higher scores indicate better patient satisfaction.
HCAHPS Communication with Nurses Composite Score | At hospital discharge (assessed up to 21 days after enrollment)
  HCAHPS Communication with Nurses composite includes 3 items rated on a 4-point frequency scale (Never/Sometimes/Usually/Always). Scores are converted to a 0-100 scale where higher scores indicate better nurse communication. Items assess whether nurses treated patient with courtesy/respect, listened carefully, and explained things understandably.
HCAHPS Communication with Doctors Composite Score | At hospital discharge (assessed up to 21 days after enrollment)
  HCAHPS Communication with Doctors composite includes 3 items rated on a 4-point frequency scale (Never/Sometimes/Usually/Always). Scores are converted to a 0-100 scale where higher scores indicate better doctor communication. Items assess whether doctors treated patient with courtesy/respect, listened carefully, and explained things understandably.
Pittsburgh Sleep Quality Index (PSQI) Global Score | Baseline, Day 2 post-enrollment, and 24 hours before procedure (assessed up to 14 days after enrollment)
  The Pittsburgh Sleep Quality Index (PSQI) assesses sleep quality over the previous night. Global score ranges from 0 to 21, with higher scores indicating worse sleep quality. A global score >5 indicates poor sleep quality.
Procedural Pain/Discomfort Visual Analog Scale (VAS) | Within 30 minutes after endoscopy procedure completion
  Visual Analog Scale (VAS) for procedural pain and discomfort ranges from 0 to 10, where 0 = no pain/discomfort and 10 = worst imaginable pain/discomfort. Higher scores indicate worse pain/discomfort. Assessed immediately post-procedure.
Total Sedation Medication Dose (Midazolam Equivalents) | During endoscopy procedure (assessed up to 14 days after enrollment)
  Total sedation medication dose administered during endoscopy, calculated as midazolam equivalents in milligrams (mg). Conversion formula: midazolam (mg) + propofol (mg)/20 + fentanyl (mcg)/100. Lower doses indicate less sedation requirement.
Endoscopy Procedure Duration | Measured intraoperatively from endoscope insertion to withdrawal; endoscopy procedure occurs within 14 days of enrollment
  Total procedure time in minutes, measured from endoscope insertion to withdrawal. Shorter duration may indicate better patient tolerance and cooperation.
Incidence of Peri-procedural Adverse Events | From procedure start through 24 hours post-procedure (assessed up to 15 days after enrollment)
  Number of participants experiencing adverse events during or within 24 hours post-procedure, graded by American Society for Gastrointestinal Endoscopy (ASGE) severity classification: mild (requires observation only), moderate (requires medical intervention), severe (requires hospitalization or ICU admission), or fatal. Events include cardiopulmonary complications (hypoxia, hypotension, arrhythmia), perforation, bleeding, aspiration, or other complications.
Hospital Length of Stay | From hospital admission to discharge (assessed up to 28 days)
  Total hospital length of stay measured in days from admission to discharge. Shorter length of stay indicates more efficient care and potentially fewer complications.
30-Day Unplanned Hospital Readmission Rate | From hospital discharge through 30 days post-discharge
  Proportion of participants with unplanned hospital readmission related to the index endoscopy procedure or its complications within 30 days of hospital discharge. Lower rates indicate better outcomes and care quality.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Lanzhou University, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] HAMILTON M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32(1):50-5. doi: 10.1111/j.2044-8341.1959.tb00467.x. No abstract available. PMID 13638508